CLINICAL TRIAL: NCT06004453
Title: Characterizing Guideline Adoption and Treatment Quality in Clinical Routine of German HFrEF Care in Heart Failure Units and Independent Centers Utilizing Established Quality Indicators
Brief Title: Characterizing Guideline Adoption and Treatment Quality in Clinical Routine of German HFrEF Care
Acronym: CONNECT
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CLCZ696BDE06
Record Dates: First submitted 2023-08-17; First posted 2023-08-22 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Heart Failure
Keywords: Heart Failure; HFrEF; patient management; quality of care; quality indicators
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other

GROUPS / COHORTS (5):
- Cohort A: Supra-regional HFU Centers and HFU Focus Hospitals
  Interventions: Other: Heart Failure medications
- Cohort B: Non-HFU Hospitals
  Interventions: Other: Heart Failure medications
- Cohort C: HFU Residential Cardiologists
  Interventions: Other: Heart Failure medications
- Cohort D: Non-HFU Residential Cardiologists
  Interventions: Other: Heart Failure medications
- Cohort E: General practitioners
  Interventions: Other: Heart Failure medications

INTERVENTIONS:
Other: Heart Failure medications — There was no treatment allocation. Patients were allocated to the respective cohort based on the treating physician enrolling them in the study. Patients were treated according to the local prescribing information and routine medical practice.

SUMMARY:
This was a multicenter, non-randomized, non-interventional cohort study with prospective and retrospective collection of primary data on heart failure with reduced ejection fraction (HFrEF) patient treatment and care following a decompensation event in different types of Heart Failure Unit (HFU) or non-HFU centers across Germany.

DETAILED DESCRIPTION:
This study aimed to describe quality of care of HFrEF patients following a decompensation event in different center types (=settings) utilizing the quality indicators for the care and outcomes of adults with heart failure as specified by the Heart Failure Association in 2022.

No strict visit schedule was imposed on participants to avoid interference with routine clinical care. HFrEF patients were treated according to the local routine in terms of medication, visit frequency and types of assessments performed and only these data was collected as part of the study from patient files.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who provide written informed consent to participate in the study
2. Male or female patients ≥ 18 years of age
3. Patients with diagnosis of heart failure with reduced ejection fraction (HFrEF) and HF treatment according to the summaries of product characteristics (SmPCs)
4. Decompensation event up to three months prior to inclusion

Exclusion Criteria:

1. Simultaneous or planned participation in an interventional research study
2. Participation in this study at another site e.g. in a HFU network
3. Patients incapable of understanding and signing the informed consent form

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Heart failure with reduced ejection fraction patients with a recent decompensation event
Sampling Method: Non-Probability Sample
Enrollment: 899 (Actual)
Dates: Start 2023-04-03 (Actual); Primary Completion 2025-01-17 (Actual); Study Completion 2025-01-17 (Actual)

PRIMARY OUTCOMES:
Quality of care and guideline adoption score in different structural settings as assessed by an opportunity-based quality indicator (QI) composite endpoint | 6 months
  Quality of care and guideline adoption score in different structural settings as assessed by an opportunity-based QI composite endpoint defined by the number of times each of secondary endpoints has been accomplished divided by chances to accomplish them as average per center type.
  To describe the quality of Heart Failure (HF) patient care in Heart Failure Unit (HFU) and non-HFU centers utilizing QIs as suggested by the 2021 European Society of Cardiology HF guideline.

SECONDARY OUTCOMES:
Proportion of sites with a dedicated multidisciplinary team to manage patients with HF | Baseline
  To describe the structural framework of the participating centers.
Percentage of sites with dedicated trained healthcare professionals to deliver HF specific education to facilitate patient self-care. | Baseline
  To describe the structural framework of the participating centers.
(A) Proportion of patients with HF who have a documentation of their HF clinical type | Baseline
  HF clinical type: Heart failure with reduced ejection fraction (HFrEF), HF with a midrange ejection fraction (HFmrEF), HF with preserved ejection fraction (HFpEF).
  To describe the patient assessment in different types of HFU and non-HFU centers.
(B) Proportion of patients with a documentation of their electrocardiogram findings | 6 months
  To describe the patient assessment in different types of HFU and non-HFU centers.
(C) Proportion of patients who have their natriuretic peptides (NPs) measured (within a 3-month period from the time of decompensation) | 3 months
  To describe the patient assessment in different types of HFU and non-HFU centers.
(D) Proportion of patients who have their blood tests documented | 3 months
  To describe the patient assessment in different types of HFU and non-HFU centers.
(E) Proportion of patients hospitalized with HF who have been referred for a cardiac rehabilitation program | 6 months
  To describe the patient assessment in different types of HFU and non-HFU centers.
(F) Proportion of patients hospitalized with HF who have a follow-up review by a healthcare professional within 4 weeks of hospital discharge | 4 weeks
  To describe the patient assessment in different types of HFU and non-HFU centers.
(G) Proportion of patients treated with beta-blocker bisoprolol, carvedilol, sustained-release metoprolol succinate, or nebivolol in the absence of any contraindications as defined by Aktaa et al 2022 | 6 months
  To describe the initial treatment algorithm of HFrEF patients following a decompensation in different types of HFU and non-HFU centers.
(H) Proportion of patients treated with an Angiotensin-converting enzymes (ACE) inhibitor, Angiotensin receptor blocker (ARB) or Angiotensin receptor-neprilysin inhibitor (ARNI) in the absence of any contraindications | 6 months
  To describe the initial treatment algorithm of HFrEF patients following a decompensation in different types of HFU and non-HFU centers.
(I) Proportion of patients treated with an Mineralocorticoid receptor antagonist (MRA) in the absence of any contraindications | 6 months
  To describe the initial treatment algorithm of HFrEF patients following a decompensation in different types of HFU and non-HFU centers.
(J) Proportion of patients treated with a Sodium-glucose co-transporter 2 (SGLT2) inhibitor in the absence of any contraindications | 6 months
  To describe the initial treatment algorithm of HFrEF patients following a decompensation in different types of HFU and non-HFU centers.
Proportion of patients receiving ARNI instead of ACEi/ARB as first-line treatment | 6 months
  To describe the initial treatment algorithm of HFrEF patients following a decompensation in different types of HFU and non-HFU centers.
Proportion of patients with HF who are prescribed loop diuretic therapy if they have evidence of fluid retention | 6 months
  To describe the initial treatment algorithm of HFrEF patients following a decompensation in different types of HFU and non-HFU centers.
Time to treatment of the above 4 individual treatment classes and time to treatment with all four classes together | 6 months
  To describe the initial treatment algorithm of HFrEF patients following a decompensation in different types of HFU and non-HFU centers.
Percentage of days covered with all four treatment classes | 6 months
  To describe the initial treatment algorithm of HFrEF patients following a decompensation in different types of HFU and non-HFU centers.
(K) Proportion of symptomatic patients with HFrEF in sinus rhythm with a QRS duration ≥150ms and left bundle branch block QRS morphology and with LVEF ≤35% despite ≥3 months optimal medical therapy who are offered cardiac resynchronization therapy | 6 months
  To describe the therapy optimization in different types of HFU and non-HFU centers.
(L) Proportion of symptomatic patients with HF, LVEF ≤35% despite ≥3 months of optimal medical therapy, and ischemic heart disease (IHD) who are offered primary prevention implantable cardioverter defibrillator | 6 months
  To describe the therapy optimization in different types of HFU and non-HFU centers.
Proportion of patients who have an assessment of their Health-related quality of life (HRQoL) using a validated tool | 6 months
  To describe the utilization of HRQoL assessments in different types of HFU and non-HFU centers.
Number of patients who are eligible for and have accomplished secondary endpoint g-j divided by the number of patients who are eligible for g-j | 6 months
  To describe quality of treatment utilizing an all-or-none composite QI.
Number of HF hospitalizations, stratified by bed type | 6 months
  Where a patient had multiple HF hospitalization stays, each hospitalization was counted.
  To describe healthcare resource utilization in patients hospitalized with HF during 6 months follow-up.
Length of hospital stay | 6 months
  Length of hospital stay was considered as the time from admission date until discharge for each HF hospitalization.
  To describe healthcare resource utilization in patients hospitalized with HF during 6 months follow-up.
Number of HF hospitalizations per patient | 6 months
  To describe healthcare resource utilization in patients hospitalized with HF during 6 months follow-up.
Number of newly implanted devices | 6 months
  implanted devices: implantable cardioverter defibrillator (ICD), Cardiac resynchronization therapy (CRT), combination of ICD and CRT (CRT-D).
  To describe healthcare resource utilization in patients hospitalized with HF during 6 months follow-up.
Number of valve interventions | 6 months
  To describe healthcare resource utilization in patients hospitalized with HF during 6 months follow-up.
Number of participants with medical history of selected comorbidities | Baseline
  To describe the HFrEF patient population with a recent decompensation

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (88):
- Germany (88):
  - Novartis Investigative Site, Heidelberg, Baden-Wurttemberg
  - Novartis Investigative Site, Ludwigsburg, Baden-Wurttemberg
  - Novartis Investigative Site, Muellheim Im Markgraeflerland, Baden-Wurttemberg
  - Novartis Investigative Site, Frankfurt am Main, Hesse
  - Novartis Investigative Site, Kassel, Hesse
  - Novartis Investigative Site, Braunschweig, Lower Saxony
  - Novartis Investigative Site, Winsen, Lower Saxony
  - Novartis Investigative Site, Löhne, North Rhine-Westphalia
  - Novartis Investigative Site, Frankenthal, Rhineland-Palatinate
  - Novartis Investigative Site, Ingelheim, Rhineland-Palatinate
  - Novartis Investigative Site, Kaiserslautern, Rhineland-Palatinate
  - Novartis Investigative Site, Kleinblittersdorf, Saarland
  - Novartis Investigative Site, Chemnitz, Saxony
  - Novartis Investigative Site, Leipzig, Saxony
  - Novartis Investigative Site, Limbach-Oberfrohna, Saxony
  - Novartis Investigative Site, Pirna, Saxony
  - Novartis Investigative Site, Halle, Saxony-Anhalt
  - Novartis Investigative Site, Jerichow, Saxony-Anhalt
  - Novartis Investigative Site, Berlin, State of Berlin
  - Novartis Investigative Site, Gera, Thuringia
  - Novartis Investigative Site, Aichach
  - Novartis Investigative Site, Amberg
  - Novartis Investigative Site, Bad Homburg
  - Novartis Investigative Site, Bad Neustadt an der Saale
  - Novartis Investigative Site, Bad Vilbel
  - Novartis Investigative Site, Bechhofen
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Bexbach
  - Novartis Investigative Site, Biedenkopf
  - Novartis Investigative Site, Bitterfeld-Wolfen
  - Novartis Investigative Site, Breuberg
  - Novartis Investigative Site, Brilon
  - Novartis Investigative Site, Bruchsal
  - Novartis Investigative Site, Brüel
  - Novartis Investigative Site, Coburg
  - Novartis Investigative Site, Coswig
  - Novartis Investigative Site, Dessau
  - Novartis Investigative Site, Dinkelsbühl
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, Düsseldorf
  - Novartis Investigative Site, Ehingen
  - Novartis Investigative Site, Erfurt
  - Novartis Investigative Site, Farchant
  - Novartis Investigative Site, Freiberg
  - Novartis Investigative Site, Fulda
  - Novartis Investigative Site, Giengen an der Brenz
  - Novartis Investigative Site, Göppingen
  - Novartis Investigative Site, Hagen
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Heidelberg
  - Novartis Investigative Site, Homburg
  - Novartis Investigative Site, Hoppegarten
  - Novartis Investigative Site, Kiel
  - Novartis Investigative Site, Kitzingen
  - Novartis Investigative Site, Kleve
  - Novartis Investigative Site, Leipzig
  - Novartis Investigative Site, Ludwigshafen
  - Novartis Investigative Site, Lübeck
  - Novartis Investigative Site, Magdeburg
  - Novartis Investigative Site, Markkleeberg
  - Novartis Investigative Site, Moers
  - Novartis Investigative Site, Münster
  - Novartis Investigative Site, Osnabrück
  - Novartis Investigative Site, Papenburg
  - Novartis Investigative Site, Potsdam
  - Novartis Investigative Site, Radebeul
  - Novartis Investigative Site, Rastatt
  - Novartis Investigative Site, Remscheid
  - Novartis Investigative Site, Rostock
  - Novartis Investigative Site, Rotenburg an der Fulda
  - Novartis Investigative Site, Rudersberg
  - Novartis Investigative Site, Schönebeck
  - Novartis Investigative Site, Schwandorf in Bayern
  - Novartis Investigative Site, Siegen
  - Novartis Investigative Site, Speyer
  - Novartis Investigative Site, Stadtlohn
  - Novartis Investigative Site, Stahnsdorf
  - Novartis Investigative Site, Stuttgart
  - Novartis Investigative Site, Ulm
  - Novartis Investigative Site, Urbach
  - Novartis Investigative Site, Wedemark
  - Novartis Investigative Site, Wermsdorf
  - Novartis Investigative Site, Wiesbaden
  - Novartis Investigative Site, Winsen
  - Novartis Investigative Site, Wismar
  - Novartis Investigative Site, Wittenberg
  - Novartis Investigative Site, Wolfsburg
  - Novartis Investigative Site, Würzburg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Link to study results — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=18384